CLINICAL TRIAL: NCT05300789
Title: Peritoneal Recurrence Among pT4 Colon Cancer Tumors: Epidemiology, Oncologic Outcomes and Risk-stratification Model. Results From an Observational Retrospective Multicenter Long-term Follow-up Study
Brief Title: Metachonous Peritoneal Carcinomatosis Incidence After Curative Surgery for pT4 Colon Cancer Patients
Status: Completed | Type: Observational
Sponsor: Carlos Cerdán Santacruz (Other)
Collaborators: Spanish Association of Surgeons (AEC) (Other)
Responsible Party: Sponsor-Investigator, Carlos Cerdán Santacruz, Consultant. Colorectal Surgery Department. Principal Investigator, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Other Study IDs: 04/21-4398
Record Dates: First submitted 2022-03-09; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Peritoneal Carcinomatosis; Colon Cancer
Keywords: colon cancer; metachronous peritoneal carcinomatosis; epidemiology; risk factors
MeSH Terms: conditions — Peritoneal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pT4 colon cancer patients after curative resection
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — There is no intervention. Patients are just going to be registered and oncologic follow-up data are going to be recorded.

SUMMARY:
This is an observational retrospective cohort study to determine metachronous peritoneal carcinomatosis in a specific subgroup of colon cancer patients, those with a final pathologic exam corresponding to pT4 tumors.

Based on a sample size calculation of 1152 patients, a retrospective review of a three year period of every participant hospitals, 50 in total, of different characteristics, was stablished.

Demographic, clinical, operative, histologic and oncologic follow-up variables were recorded.

DETAILED DESCRIPTION:
This is an observational retrospective cohort study to determine metachronous peritoneal carcinomatosis in a specific subgroup of colon cancer patients, those with a final pathologic exam corresponding to pT4 tumors.

A national multicenter retrospective cohort study is proposed. Given that the objectives of the study is to establish the prognostic oncologic impact of developing metachronous peritoneal carcinomatosis, it is intended to include patients who have completed three years of follow-up, therefore, the period of inclusion of patients to be analyzed is from 2015 to 2017.

Inclusion criteria:

* Patients operated on for colon cancer, considering those patients with neoplasia located from 15 cm from the anal margin in the proximal direction.
* Patients with histological confirmation of colon adenocarcinoma.
* Postoperative anatomical-pathological staging pT4a and pT4b.
* Patients operated both electively and urgently.
* Patients in whom a complete macroscopic resection of the primary tumor is achieved.

Exclusion criteria:

* Histological types other than adenocarcinoma, such as leiomyosarcomas, GIST, neuroendocrine tumors and other less frequent forms.
* Patients in whom the persistence of macroscopic oncological disease is described after the intervention on the primary tumor, considering it totally unresectable.

Definitions:

Definition of peritoneal carcinomatosis: presence of oncological disease at the peritoneal level, whether single or multifocal, and that is clearly recognizable and distinguishable from other forms of loco-regional recurrence of colon cancer such as anastomotic, mesenteric or lymph node recurrence and retroperitoneal form.

Definition of second look type surgery: it is considered all that programmed intervention carried out to rule out the presence of peritoneal carcinomatosis based on anatomo-pathological or clinical data related to the primary tumor and its debut form, but without the existence of clinical, analytical data or radiological during follow-up that allow it to be suspected.

Variables collected:

* Center code: each participating center will receive an exclusive code that will be the first variable in the database in order to identify the participation of each center in the study.
* Patient code: each patient included in each center will receive a consecutive numerical code to identify the participation of each center in the study.
* Demographic variables: sex, date of birth, body mass index (BMI).
* Patient comorbidity: the comorbidity of the collected patients will be shown exclusively with the anesthetic risk of the American Association of Anesthesiology (ASA Score).
* Primary neoplasm: diagnosis by presence and type of symptoms or diagnosis in the asymptomatic phase, location of the tumor and preoperative clinical staging based on extension studies.
* Operative data: date of the intervention, type of intervention (urgent vs. scheduled), approach, findings, type of resection performed, primary anastomosis or not, diverting or terminal stoma and postoperative complications at 30 days, especially those of infectious origin intra-abdominal. The rest of the complications that arise will be collected according to the Clavien-Dindo classification but will not be specified.
* Anatomical-pathological data: result of the cytological study if it has been carried out, histological type of the tumor, degree of differentiation, tumor staging according to the TNM classification and other histological prognostic criteria such as vascular, lymphatic and perineural infiltration.
* Adjuvant treatments: it will be collected if the patient underwent adjuvant treatment or not and if the proposed chemotherapy scheme could be carried out completely or was interrupted for any reason.
* Follow-up: performance of second look type surgery, findings during it, surgical technique performed, appearance or not of recurrence and the date of recurrence, type of recurrence (peritoneal carcinomatosis or distant metastasis), form of diagnosis of recurrence ( clinical, analytical, radiological or histological confirmation), salvage surgery for peritoneal carcinomatosis and, if so, rate of peritoneal carcinomatosis and technique used, performed in the same center or referral of the patient, performed by a unit specialized in surgery of peritoneal carcinomatosis or not, mortality and whether this was caused by the terminal evolution of the oncological process and the date of the last control (date of death or date of the last follow-up of the patient), with which the disease-free survival and the overall survival.

Calculation of the sample size. To carry out an adequate calculation of the sample size, the only multicenter prospective study at the national level of patients operated on for colon cancer, the ANACO study, has been used as a reference. In that study, with 52 participating centers, during a full year 3230 patients were registered who, after applying different exclusion criteria, remained in 2968, of which 550 patients were classified as T4 tumors after the histological study, that is, almost 20% of the tumors operated on in our environment.

Based on these figures, assuming a degree of participation similar to that obtained in the ANACO study, establishing an approximate figure of 1,500 pT4a/b colon tumors as the target population over the three years of study in our country. , an incidence of peritoneal carcinomatosis of approximately 15%, a confidence level of 95% and a precision of +/- 1 percentage units, a random sample of 1152 individuals is sufficient for the estimate to be made in this work.

Statistical method A descriptive analysis of demographic and clinical variables will be performed. Categorical variables will be presented as percentages and frequencies. The distribution of continuous variables will be evaluated using the Shapiro-Wilk statistic and they will be described as mean and standard deviation if they follow a normal distribution or as median and interquartile range (IQR) otherwise.

The association between the variables collected and the objective variables of the study will be made using Pearson's Chi-square test or Fisher's exact test, as appropriate, in the case of categorical variables and, for continuous variables, using Student's t-test for independent samples or Mann-Whitney U, respectively, depending on whether or not their distribution is adjusted to normal.

Project schedule and phases

* November - December 2020: Preparation and approval of the study protocol by the members of the Coloproctology Section of the Spanish Association of Surgeons.
* January - February 2020:

  * Application for approval by the local ethics committees of the centers of the members of the Section involved in the project.
  * Invitation to participate in the study by means of a formal letter to the department heads of the centers considered most representative and with the greatest volume in colon cancer surgery. For this purpose, the registry of participating centers in the previous ANACO registry has been used.
  * Open invitation to all members of the Spanish Association of Surgeons through official communication by the Section of the start-up of the study.
  * Preparation of the database in Excel format for later dissemination among the study participants.
* March - June 2020:

  * Confirmation and commitment by the centers interested in participating in the study.
  * Collection of data and sending of the files to those responsible for the project.
* July September:

  * Condensation of the data from the different files into a single file.
  * Statistical study and obtaining results.
* October - December 2021:

  * Preparation of an original manuscript for submission and assessment for publication.

ELIGIBILITY:
Inclusion Criteria:

* Colon cancer above 15 cm from anal verge
* Curative intent surgery
* Pathologic confirmation of pT4 adenocarcinoma

Exclusion Criteria:

* R2 cancer resection
* Inclusion in other randomized clinical trials
* Pathologic diagnosis of colon cancer other than adenocarcinoma, such as GIST, leiomyosarcomas, neuroendocrine tumors, or other types even more unusual.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult colon cancer patients operated on with curative intention, both scheduled and emergency surgery, with pathologic confirmation of pT4 tumors.
Sampling Method: Non-Probability Sample
Enrollment: 1152 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Metachronous peritoneal carcinomatosis | A minimum of 3-years follow-up
  Number of patients diagnosed with peritoneal carcinomatosis during regular oncologic follow-up

SECONDARY OUTCOMES:
Time to metachronous peritoneal carcinomatosis diagnosis | A minimum of 3-years follow-up
  Time (months) from surgical treatment of primary tumor to diagnosis of peritoneal carcinomatosis during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Carlos Cerdán, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All information regarding this study will be shared under demand and with well documented and reasonable arguments.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From the present moment, during the next 3 years.
Access Criteria: Under demand and with well documented and reasonable arguments.